CLINICAL TRIAL: NCT00217568
Title: A Phase II Trial of Docetaxel and Carboplatin for First Relapsed Platinum-Sensitive Stage III and IV Advanced Ovarian Cancer or Peritoneal Carcinoma
Brief Title: Docetaxel and Carboplatin in Treating Patients With Relapsed Stage III or Stage IV Ovarian Epithelial or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: PSOC 1702; PSOC-1702; AVENTIS-PSOC-1702; PSOC-IRB-4861; CDR0000441307 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — pegfilgrastim; Carboplatin; Docetaxel

INTERVENTIONS:
Biological: pegfilgrastim
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with carboplatin works in treating patients with relapsed stage III or stage IV ovarian epithelial or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of docetaxel and carboplatin in patients with platinum-sensitive stage III or IV ovarian epithelial or primary peritoneal cavity cancer in first relapse.
* Determine the response rates (complete and partial response) in patients treated with this regimen.
* Determine relapse rates and event-free survival and overall survival rates in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Patients also receive pegfilgrastim subcutaneously on day 2 . Treatment repeats every 21 days for up to 6 courses.

After completion of study treatment, patients are followed at 3 weeks, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal cavity cancer

  * Stage III or IV disease
  * No borderline tumors
* Measurable or evaluable disease

  * Measurable disease, defined as evidence of disease by physical examination or radiographic evaluation
  * Evaluable disease, defined as CA 125 ≥ 100 U/mL (confirmed by 2 blood tests performed ≥ 1 week apart)
* In first relapse

  * Platinum-sensitive disease, defined as initial relapse > 6 months after completion of a platinum-based regimen

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * SGOT and/or SGPT ≤ 1.5 times upper limit of normal (ULN) AND alkaline phosphatase (AP) ≤ 2.5 times ULN
  * SGOT and/or SGPT ≤ 5.0 times ULN AND AP normal

Renal

* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance > 50 mL/min

Cardiovascular

* LVEF ≥ 50%
* No poorly controlled arrhythmia
* No unstable coronary artery disease or myocardial infarction within the past year

Other

* HIV negative
* No pre-existing peripheral neuropathy > grade 2
* No history of allergy to study drugs

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy and recovered

Surgery

* Recovered from recent prior surgery

Other

* No concurrent myelosuppressive therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-05; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Toxicity
Response rates (complete and partial response)
Relapse rates
Event-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington